CLINICAL TRIAL: NCT03331679
Title: Exploring Time Efficient Strategies to Improve Fitness for Surgery in Older Adults- Two Weeks HIIT
Brief Title: Can 2 Weeks of High Intensity Interval Training in Healthy 65-85 Year-olds Improve Cardiorespiratory Fitness?
Acronym: 2WkHIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A12092016 amendment 4
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Cardiorespiratory Fitness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 2 Wk HIIT (Experimental): 2 weeks of High Intensity Interval Training
  Interventions: Behavioral: HIIT

INTERVENTIONS:
Behavioral: HIIT — 2 Weeks of High Intensity Interval Training on a Cycle ergometer

SUMMARY:
The incidence of conditions requiring surgical intervention increases with age, however there is a reported decline in the rates of elective surgical procedures in those over 65. This is associated with older patients being described as "less fit" and more at risk of postoperative complications, leading to decreased provision of surgical care to those at need. Exercise interventions have the potential to reverse some of the decline in cardiovascular fitness associated with aging and improve the elderly's' "fitness for surgery" and potentially allow increased access to surgical care for those most in need of it.

DETAILED DESCRIPTION:
The percentage of people aged >65 y in the United Kingdom increased from 15% in 1985 to 17% in 2010, an increase of 1.7 million people. One age-associated physiological change is the reduction in vascular function that is observed, both at the levels of the large arteries and the muscle microvasculature. In itself this vascular dysfunction is associated with reduced aerobic performance. Cardiorespiratory fitness (marked by aerobic performance) has been shown to be an independent predictor of postoperative mortality, which provides more accurate prognostic information than age alone. In contrast, physical activity can reverse elements of pathophysiology associated with these conditions, including vascular dysfunction. Nonetheless, major roadblocks to exercise as a strategy to combat age-associated vascular dysfunction and associated conditions exist, such as poor exercise tolerance and "lack of time".

The aim of this study is to investigate whether if novel low-volume, time-efficient training strategies can improve indices of vascular health and cardiorespiratory performance in older individuals with a view towards improving their fitness for surgery. Numerous studies have demonstrated that periods of supervised exercise training effectively improve indices of cardiorespiratory (blood pressure, aerobic capacity and blood lipids and vascular function. However, the majority of these studies were conducted using high-volume continuous submaximal aerobic training (e.g. 50-65% VO2max for 30-60 min) or moderate to high volume progressive weight training. This research group have recently shown the efficacy of a time-efficient exercise strategy known as HIIT - High Intensity Interval Training, for improving VO2 max and muscle mass in young individuals with heightened metabolic disease risk and also demonstrated significant improvements in VO2 max comparable to classic aerobic exercise training using several different time-efficient HIIT protocols in as little as 4 weeks. This study aims to quantify the benefits of 2 weeks of HIIT.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer aged 65-85

Exclusion Criteria:

* Current participation in a formal exercise regime
* BMI < 18 or > 32 kg·m2
* Active cardiovascular disease:
* uncontrolled hypertension (BP > 160/100),
* angina,
* heart failure (class III/IV),
* Significant arrhythmia,
* right to left cardiac shunt,
* recent cardiac event
* Taking beta-adrenergic blocking agents,
* Cerebrovascular disease: previous stroke, aneurysm (large vessel or intracranial)
* epilepsy
* Respiratory disease including: pulmonary hypertension, Significant COPD, Uncontrolled asthma, Metabolic disease: -hyper and hypo parathyroidism, -untreated hyper and hypothyroidism, Cushing's disease, type 1 or 2 diabetes
* Active inflammatory bowel or renal disease
* Malignancy
* Clotting dysfunction
* Significant Musculoskeletal or neurological disorders
* Family history of early (<55y) death from cardiovascular disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Anaerobic Threshold | 2 weeks
  Anaerobic Threshold as measured at standard CPET conducted according to ATS/ACCP statement (measured in ml/Kg/min)

SECONDARY OUTCOMES:
VO2 Peak | 2 Weeks
  Maximum volume of oxygen consumed at CPET conducted according to ATS/ACCP statement (measured in ml/Kg/min)
Whole-Body Lean Mass | 2 Weeks
  Measured by DEXA (Kg)
Body Fat percentage | 2 Weeks
  Measured by DEXA
Leg Lean Mass | 2 Weeks
  Measured by DEXA (Kg)
Handgrip Strength | 2 Weeks
  Maximum voluntary contraction

CONTACTS AND LOCATIONS:
Locations (1):
- Medical School, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided